CLINICAL TRIAL: NCT06435715
Title: The Effect of 10 Repetitions of Deep Breathing Exercises Compared to 3 Repetitions of Deep Breathing Exercises on The Sleep Quality of Post-Cardiac Surgery Patients
Brief Title: The Effect of 10 Repetitions of Deep Breathing Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Indra Gilang Pamungkas, Ns. Indra Gilang Pamungkas, S.Kep., M.Kep, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DP.04.03/KEP071/EC027/2024
Record Dates: First submitted 2024-05-26; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result
Keywords: Breathing Exercise; Sleep Quality; Cardiac Surgical Procedures
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study used a parallel Randomized Controlled Trial (RCT) with a 1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were not involved during the intervention process. Respondents were also asked not to inform the outcome assessor of the measures they received.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The group that carries out the intervention of the treatment being studied
  Interventions: Other: 10 Repetitions of Deep Breathing Exercise
- Control Group (Active Comparator): The group that did usual care
  Interventions: Other: 3 Repetitions of Deep Breathing Exercise

INTERVENTIONS:
Other: 10 Repetitions of Deep Breathing Exercise — Respondents in the intervention group performed 10 repetitions of deep breathing exercises every 3 hours for 3 days.
  Arms: Intervention Group
Other: 3 Repetitions of Deep Breathing Exercise — Respondents in the control group performed 3 repetitions of deep breathing exercises for 3 days.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn and assess the effect of 10 repetitions of deep breathing exercises every 3 hours compared to 3 repetitions of deep breathing exercises on the sleep quality of patients after heart surgery.

The main questions it aims to answer are:

How does 10 repetitions of deep breathing exercises every 3 hours affect the sleep quality of patients after heart surgery?

Researchers will compare 10 repetitions of deep breathing exercises every 3 hours to 3 repetitions of deep breathing exercises to see if 10 repetitions of deep breathing exercises every 3 hours work to improve sleep quality.

Participants will:

1. Respondents in the intervention group performed 10 repetitions of deep breathing exercises every 3 hours for 3 days.
2. Respondents in the control group performed 3 repetitions of deep breathing exercises for 3 days.

DETAILED DESCRIPTION:
1. Researchers carried out recruitment when the patient had undergone surgery.
2. Researchers determine potential respondents who meet the inclusion criteria.
3. Researchers explain to potential respondents the procedures, objectives, benefits and risks of the research being conducted.
4. Researchers provide time and opportunity for potential respondents to confirm research procedures.
5. The researcher provided an informed consent sheet as a form of respondent's agreement to their involvement in the research.
6. Researchers determine respondents for the intervention and control groups.
7. Respondents do a pretest. The pretest was administered by administering a sleep characteristics and quality questionnaire.
8. Researchers provide education to patients regarding deep breathing exercise procedures.
9. Respondents in the intervention group performed deep breathing exercises with 10 repetitions every 3 hours for 3 days. Respondents in the control group did 3 repetitions of deep breathing exercises.
10. Respondents are monitored in the implementation process using a monitoring form.
11. Respondents who completed the exercise will conduct a post-test assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone cardiac surgery, both on-pump and off-pump.
* The patient's hemodynamic condition is stable.
* More than equal to 18 years old.
* Able to communicate, read and write in Indonesian.

Exclusion Criteria:

* Patients who receive sleeping medication or sedative therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | 30 minutes
  Sleep quality experienced by patients after undergoing heart surgery

CONTACTS AND LOCATIONS:
Overall Officials: Indra G Pamungkas, Master, Study Chair — Indonesia University
Locations (1):
- National Cardiovascular Centre Harapan Kita, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Result] Ghorbani A, Hajizadeh F, Sheykhi MR, Mohammad Poor Asl A. The Effects of Deep-Breathing Exercises on Postoperative Sleep Duration and Quality in Patients Undergoing Coronary Artery Bypass Graft (CABG): a Randomized Clinical Trial. J Caring Sci. 2018 Dec 1;8(4):219-224. doi: 10.15171/jcs.2019.031. eCollection 2019 Dec. PMID 31915624